CLINICAL TRIAL: NCT04075279
Title: Cardiovascular Mechanisms of the Occupational Physical Activity Health Paradox: 24-hour Physical Activity, Blood Pressure, and Heart Rate
Brief Title: Heart at Work Study
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Tyler Quinn, Principle Investigator, University of Pittsburgh
Other Study IDs: STUDY19050097
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Occupational Diseases; Cardiovascular Diseases; Cardiovascular Risk Factor; Occupational Exposure
MeSH Terms: conditions — Occupational Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to examine the cardiovascular mechanisms of increased cardiovascular mortality in those with high activity occupations.

DETAILED DESCRIPTION:
The current proposal uses a repeated-measures, within-subject design to address our aims. Twenty male participants will report to the laboratory to provide informed consent, complete baseline assessments, and receive ambulatory monitors. Following this session, each participant will wear physical activity and ambulatory cardiovascular monitors for 7 days, including at least one non-work day and one work day. Characterization of work activity will use physical activity data from self-reported time at work (Specific Aim I). The 24-hour cardiovascular load (HR and BP) and nocturnal HRV will be compared across work and non-work days (Specific Aim II). Lastly, whether fitness level or job strain modify the difference in cardiovascular strain between work vs. non-work days will be evaluated (Specific Aim III).

ELIGIBILITY:
Inclusion Criteria:

* middle age (35-59 years)
* male
* self-report working full-time in the food service industry (≥30 hours/week)
* self-report predominantly completing light intensity activity job responsibilities (≥75% work time walking, light movement, or standing)

Exclusion Criteria:

* Resting blood pressure of ≥150 mmHg systolic and/or ≥95 mmHg diastolic
* currently taking medications that are known to affect blood pressure or heart rate (e.g. Beta-blockers, ACE inhibitors, etc.)
* greater than low risk to participate in physical activity as determined by PAR-Q (answer of yes to any of the 7 physical activity readiness questionnaire questions)
* report working a second job in addition to their primary full-time job
* report working overnight shifts (10pm-6am)
* reported physical dysfunction (inability to walk 2 city blocks or climb 2 flights of stairs)
* inability to complete the sub-maximal exercise test to completion (80% age-predicted heart rate maximum)
* Currently being treated for a serious medical condition such as kidney disease, liver disease, cancer, or heart disease.

Ages: 35 Years to 59 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes — Only males are eligible for this study.
Study Population: Middle-aged male food service workers
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler D Quinn, MS, Principal Investigator — Graduate Student
Locations (1):
- Physical Activity and Weight Management Research Laboratory, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Upon completion of all data collection, data will be analyzed and summary conclusions will be published in a peer reviewed scientific journal.

REFERENCES:
- [Derived] Quinn TD, Bruehwiler T, Chantler PD, Gibbs BB. Cardiovascular Responses to Occupational Physical Activity Are Exaggerated by Work-Related Stress and Low Fitness. J Occup Environ Med. 2024 Oct 1;66(10):e476-e482. doi: 10.1097/JOM.0000000000003183. Epub 2024 Jul 1. PMID 38955811

RESULTS

PARTICIPANT FLOW:
Groups:
- Middle-aged Males in High Activity Occupations: All participants were enrolled into a single arm and all comparisons were made within subjects.
Period: Overall Study
Arm/Group | Middle-aged Males in High Activity Occupations
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Research Study Participation: Participants who were enrolled in the study and completed all study procedures.
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 13
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
Occupational Industry [Count of Participants; unit: Participants]
  Food Service | 8
  Material Moving | 9
  Healthcare | 1
  Building and Grounds Maintenance | 1

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Heart Rate
Description: We will calculate the average heart rate over each 24 hour period throughout a one week monitoring period.
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
beats per minute
  Workdays | 83.8 (1.2)
  Non-workdays | 78.5 (1.4)

2. Secondary Outcome: 24-hour Ambulatory Systolic Blood Pressure
Description: We will calculate the average systolic blood pressure over a 24-hour period on two separate days (workdays versus non-workdays).
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Error); unit: millimeters of Mercury
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
millimeters of Mercury
  Workdays | 126.0 (1.7)
  Non-workdays | 124.0 (1.8)

3. Secondary Outcome: Nocturnal Heart Rate Variability, RMSSD
Description: We will calculate the average heart rate variability during each night's sleep for a total of one week. The specific HRV variable presented is root mean square successive differences (RMSSD).
Time Frame: approximately 8 hours (sleep time)
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
milliseconds
  workdays | 34.17 (4.04)
  non-workdays | 35.34 (4.32)

4. Secondary Outcome: Physical Activity Pattern. Steps Per Day
Description: This physical activity metric of steps per day was calculated as average number of steps during each day type (work versus non-workdays) throughout one week
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: steps per day
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
steps per day
  Workdays | 12,772 (945)
  Non-workdays | 7,923 (1,063)

5. Secondary Outcome: Nocturnal Heart Rate Variability, SDNN
Description: We will calculate the average heart rate variability during each night's sleep for a total of one week. The specific HRV variable presented is standard deviation of the normal to normal RR intervals (SDNN).
Time Frame: approximately 8 hours (sleep time)
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
milliseconds
  workdays | 39.85 (3.48)
  non-workdays | 42.14 (3.71)

6. Secondary Outcome: Nocturnal Heart Rate Variability, LF
Description: We will calculate the average heart rate variability during each night's sleep for a total of one week. The specific HRV variable presented is low frequency power (LF).
Time Frame: approximately 8 hours (sleep time)
Measure: Least Squares Mean (Standard Error); unit: log milliseconds
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
log milliseconds
  workdays | 6.18 (0.20)
  non-workdays | 6.45 (0.21)

7. Secondary Outcome: Nocturnal Heart Rate Variability, HF
Description: We will calculate the average heart rate variability during each night's sleep for a total of one week. The specific HRV variable presented is high frequency power (HF).
Time Frame: approximately 8 hours (sleep time)
Measure: Least Squares Mean (Standard Error); unit: log milliseconds
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
log milliseconds
  workdays | 5.22 (0.30)
  non-workdays | 5.56 (0.31)

8. Secondary Outcome: Physical Activity Pattern. MVPA
Description: This physical activity metric of minutes of moderate to vigorous physical activity was calculated as average minutes during each day type (work versus non-workdays) throughout one week
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: minutes per day
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
minutes per day
  Workdays | 72.4 (7.2)
  Non-workdays | 41.5 (8.9)

9. Secondary Outcome: Physical Activity Pattern. LPA
Description: This physical activity metric of minutes of light physical activity was calculated as average minutes during each day type (work versus non-workdays) throughout one week
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: minutes per day
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
minutes per day
  Workdays | 391.5 (19.9)
  Non-workdays | 285.2 (23.3)

10. Secondary Outcome: Physical Activity Pattern. Sedentary
Description: This physical activity metric of minutes of sedentary time was calculated as average minutes during each day type (work versus non-workdays) throughout one week
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: minutes per day
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
minutes per day
  Workdays | 492.5 (18.4)
  Non-workdays | 629.7 (22.5)

11. Secondary Outcome: Physical Activity Pattern. Upright
Description: This physical activity metric of minutes of upright time was calculated as average minutes during each day type (work versus non-workdays) throughout one week
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: minutes per day
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
minutes per day
  Workdays | 462.4 (18.4)
  Non-workdays | 325.2 (22.5)

12. Secondary Outcome: 24-hour Ambulatory Diastolic Blood Pressure
Description: We will calculate the average diastolic blood pressure over a 24-hour period on two separate days (workdays versus non-workdays).
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Error); unit: millimeters of Mercury
Arm/Group | Research Study Participation
Number analyzed (Participants) | 19
millimeters of Mercury
  Workdays | 75.2 (1.0)
  Non-workdays | 72.6 (1.1)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Research Study Participation
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT04075279/Prot_SAP_ICF_000.pdf